CLINICAL TRIAL: NCT01503385
Title: A Randomized Phase II Trial of Cisplatin/Etoposide and Concurrent Radiotherapy With or Without Celecoxib in Patients With Unresectable Locally Advanced Non-small Cell Lung Cancer
Brief Title: Cisplatin/Etoposide and Concurrent Radiotherapy With or Without Celecoxib in Patients With Unresectable Locally Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Luhua Wang, Luhua Wang, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-L-025
Record Dates: First submitted 2012-01-01; First posted 2012-01-04 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2012-01

CONDITIONS: Lung Cancer
Keywords: Celecoxib; phase II
MeSH Terms: conditions — Lung Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Celecoxib (Experimental): Combination of and concurrent radiotherapy Cisplatin/etoposide with or without Celecoxib.
  Intervention: Drug: Celecoxib
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — 400 mg by mouth twice daily for for 5-7 days before beginning radiation therapy; continued 7 days per week throughout radiation treatment (about 6 weeks).
  Other Names: Celebrex

SUMMARY:
Concurrent chemoradiation (ChRT) is a standard care for unresectable stage III non-small cell lung cancer (NSCLC) patients with good performance status, and cisplatin/etoposide (EP) regimen is one of the most commonly used regimens. However, the prognosis of these patients is still rather poor. It has been demonstrated that Cyclooxygenase (COX)-2 plays an important role in the pathogenesis of lung cancer. Selective (COX)-2 inhibitors can promote chemosensitivity and radiosensitivity of tumor cells in preclinical trials.

This is a single-institution, open-label, randomized phase II trial of celecoxib administered concurrently with cisplatin, etoposide, and radiation therapy in patients with locally advanced NSCLC, to determine the feasibility, activity, and toxicity of this combination on unresectable NSCLC, and further to examine biomarkers to predict response to the treatment.

DETAILED DESCRIPTION:
Celecoxib is a non-steroidal-anti-inflammatory drug (NSAIDS) Recent studies have shown that celecoxib has antitumor activity, and may increase the tumor sensitivity to radiation. Furthermore, evidence has shown the safety and efficiency of celecoxib in some phase I/II studies. The purposes of this study are to examine the effects of a new combination of celecoxib (Celebrex®) and cisplatin/etoposide (EP regimen), with concurrent thoracic radiotherapy on unresectable stage III NSCLC patients; and to examine biomarkers to predict response to the treatment. Because of poor survival of patients with unresected locally advanced NSCLC, the efficiency of celecoxib plus concurrent EP chemoradiotherapy need to be further investigated.

ELIGIBILITY:
Inclusion Criteria:

* • 18-70 years old, male or female

  * Histological or cytological evidence of NSCLC.
  * Unresectable Stage III NSCLC.
  * Karnofsky score: at least 70.
  * Estimated survival: at least 6 months
  * Not receiving radiotherapy or combined modality therapy to treat another malignancy.
  * No history of active gastric ulcer, active GI bleeding, or renal failure.
  * No severe hypertension, cardiac disease, or diabetes mellitus
  * Normal blood routine and chemical tests
  * Patients or guardian must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* • Other malignancies simultaneously except in situ cervix or non-melanoma skin cancer

  * Extensive distant metastases
  * Pregnancy or in lactation
  * Allergic to Sulfonamides, NSAIDS or Celebrex
  * Routine use of NSAIDS such as high dose of Aspirin
  * History of cardiovascular diseases including: myocardial infraction, angina, coronary angioplasty, congestive heart failure, stroke, or coronary bypass surgery in the last 6 months.
  * Abnormal coagulation or history of deep venous thrombosis, pulmonary embolism, systemic lupus erythematous, family history of protein S or C deficiencies, prior heparin-induced thrombocytopenia, Factor V Leiden deficiencies or high homocysteine levels.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 year overall survival

SECONDARY OUTCOMES:
progression-free survival | 3 year progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Luhua Wang, Doctor, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Jun Liang, Beijing, Beijing Municipality

REFERENCES:
- [Derived] Bi N, Liang J, Zhou Z, Chen D, Fu Z, Yang X, Feng Q, Hui Z, Xiao Z, Lv J, Wang X, Zhang T, Wang X, Deng L, Wang W, Wang J, Liu L, Hu C, Wang L. Effect of Concurrent Chemoradiation With Celecoxib vs Concurrent Chemoradiation Alone on Survival Among Patients With Non-Small Cell Lung Cancer With and Without Cyclooxygenase 2 Genetic Variants: A Phase 2 Randomized Clinical Trial. JAMA Netw Open. 2019 Dec 2;2(12):e1918070. doi: 10.1001/jamanetworkopen.2019.18070. PMID 31851351